CLINICAL TRIAL: NCT03421990
Title: Comparative Study of the Change in Liver Enzymes After General or Spinal Anesthetic Techniques in Patients With Preoperatively Elevated Liver Enzymes
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Hala Mostafa Gomaa (Unknown); Norhan Abdelaleem Ali (Unknown); Shady Abo El ela Ismaiel (Unknown); Mohamed, Ahmed A., M.D. (Individual)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia&I.C.U and Pain Clinic, Cairo University
Other Study IDs: N 30-2017/Ms
Record Dates: First submitted 2018-01-09; First posted 2018-02-05 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Liver Enzymes After General or Spinal Anesthetic Techniques; In Patients With Preoperatively Elevated Liver Enzymes
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples Without DNA — Blood Samples Liver Enzymes measurments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: General anesthesia technique
  Interventions: Procedure: General anesthesia
- Group B: Regional anesthesia technique
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: General anesthesia — general anesthesia and regional anesthesia techniques are used
  Other Names: Regional anesthesia

SUMMARY:
* To assess the changes in liver functions postoperatively in patients with preoperatively elevated liver enzymes.
* To identify the most appropriate anesthesia technique for patients with preoperatively elevated liver enzymes.
* To assess the effect of intraoperative event (bleeding, hypoxia, hypotension, prolonged operation) on liver functions in these patients.

DETAILED DESCRIPTION:
Surgery and anesthesia are stressful events, thus there is a possibility that liver enzymes and bilirubin may increase postoperatively. Mild elevations of serum aminotransferase, alkaline phosphatase, or bilirubin levels are frequent after surgical procedures, whether performed under general or spinal anesthesia. Anesthesia causes an initial reduction in hepatic arterial blood flow of 35-42% in the first 30 min of induction of anesthesia. During surgery, The liver blood flow returns to baseline. It is possible that either the initial hypoperfusion or reperfusion injury, or both, may contribute to postoperative liver dysfunction when it occurs.

The type of surgery is potentially an important factor of postoperative hepatic dysfunction. Intra-abdominal operations are more likely than extra-abdominal surgeries to cause reflex systemic hypotension and to subsequently reduce hepatic blood flow.This could be due to traction on abdominal viscera. Hypercarbia-induced splanchnic vasoconstriction is also a threat to hepatic perfusion in laparoscopic surgery. Surgeries that result in a large amount of blood loss increase the risk for ischemic hepatic injury, as can intraoperative hypotension.

Liver disease is important to recognize preoperatively because the risk of surgery in patients with advanced disease can be grave.Patients with liver disease are more likely than patients without liver disease to experience hepatic decompensation with anesthesia. Measurement of serum Bilirubin levels is central to the evaluation of hepatobiliary disorders. Liver disease is a challenging condition for the anesthesiologist, However, the risk could be diminished by careful consideration of the patients' condition preoperatively and choosing suitable anesthetic procedure and drugs for these patients.Meanwhile, The effect of performing spinal anesthesia on patients with liver disease has not been investigated properly as most studies excluded patients with preoperatively elevated liver enzymes. Studies on patients undergoing general anesthesia with normal preoperative liver function tests showed a transient increase in the level of AST& ALT, with a mild increase in postoperative bilirubin levels

ELIGIBILITY:
Inclusion Criteria:

Adult healthy ASA I, II patients, both genders, aged 18 - 60 years, with stationary elevated liver enzymes < 2 folds undergoing elective lower abdominal wall or limb surgeries with expected operation time less than 2 hours

Exclusion Criteria:

* ASA class III or IV
* Age >60 years or <18 years
* Patients undergoing intraperitoneal and laparoscopic procedures.
* Acute viral hepatitis: inflammation of the liver caused by infection with one of the five hepatitis viruses. In most people, the inflammation begins suddenly and lasts only a few weeks.
* Acute alcoholic hepatitis: is inflammation of the liver due to excessive intake of alcohol. It is usually found in association with fatty liver, an early stage of alcoholic liver disease, and may contribute to the progression of fibrosis, leading to cirrhosis.
* Severe chronic hepatitis: is inflammation of the liver that lasts at least 6 months.
* Child's C class classification: this score is used to assess the prognosis of chronic liver disease, mainly cirrhosis.
* Severe coagulopathy: a pathological condition that reduces the ability of the blood to coagulate, resulting in uncontrolled bleeding. A platelet count of < 50 x 109 /L will be considered at high risk of increased bleeding.
* Severe extrahepatic complication (Hypoxemia, Acute renal failure…)
* Pregnant, diabetic patients
* Patients having an auto-immune disease
* Patients taking anticoagulant drugs or drugs that cause elevated liver enzymes (non-steroidal anti-inflammatory drugs, antibiotics, antiepileptic drugs, inhibitors of hydroxyl-methyl-glutaryl-coenzyme a reductase (statins), and anti-tuberculosis drugs) were excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 Patients are randomly divided by computer designed lists and then concealed in closed envelopes into 2 equal groups:
  1. Group A(n=30),in which general anesthesia technique is used
  2. Group B(n=30),in which regional anesthesia technique is used
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Compare the pre and postoperative liver enzymes | 24 hours from the start
  The pre and 24 hours postoperative AST levels of patients in the general anaesthesia group and spinal anaesthesia group

SECONDARY OUTCOMES:
Changes in Liver function tests (AST, ALT, total and direct Bilirubin) from the preoperative values to 48 hours postoperative | During Operation and 48 hours postoperative
  To determine the changes in Liver function tests (AST, ALT, total and direct Bilirubin) from the preoperative values to 48 hours postoperative
Intraoperative monitoring and correlation with the change of the liver enzymes postoperative | During Operation and 48 hours postoperative
  To monitor the intraoperative vital signs (Blood pressure and Heart rate), the intraoperative blood loss and total fluid consumptions, the total consumptions of the vasopressors, the intraoperative adverse events(severe hypotension, bleeding, blood transfusion, hypoxia, hepatotoxic drugs …) and correlate it to the change of the liver enzymes postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Norhan abd Aleem Ali, M.D, Principal Investigator — Cairo University; Shady Abo El ela Ismaiel, Ph.D, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Ahmed Abdalla Mohamed, Cairo
  - Ahmed Abdalla, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
* To identify the most appropriate anesthesia technique for HCV +ve patients.
  * To assess the changes in liver functions & APRI score preoperative and postoperative in HCV +ve patients.
  * To assess the effect of intraoperative event (bleeding,hypoxia (bleeding,hypoxia,hypotension,prolonged operation )and postoperative events on liver functions in HCV +ve patients